CLINICAL TRIAL: NCT01338506
Title: Integrated Treatment of Operation Enduring Freedom/Operation Iraqi Freedom Veterans With Post-traumatic Stress Disorder and Substance Use Disorders
Brief Title: Integrated Treatment of OEF/OIF Veterans With PTSD & Substance Use Disorders
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sudie E. Back, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA030143-01 (NIH); HR20279 (Other: MUSC)
Record Dates: First submitted 2011-04-08; First posted 2011-04-19 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Posttraumatic Stress Disorders; Combat Disorders; Alcohol Dependence; Drug Dependence
Keywords: Military; Posttraumatic Stress Disorder; PTSD; PostTraumatic Stress Disorders; Combat; Psychological Treatment; Psychotherapy; Trauma; Posttraumatic Stress; Prolonged Exposure; Exposure therapy; Behavior Therapy; Cognitive Behavior Therapy; Stress Disorders; Drug Abuse; Drug Dependence; Alcohol Abuse; Alcohol Dependence; Substance Use Disorders; Alcoholism
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Alcoholism; Substance-Related Disorders; Wounds and Injuries; Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPE Therapy (Experimental): Combined prolonged exposure therapy for PTSD with cognitive behavioral therapy for substance use disorder.
  Interventions: Behavioral: Concurrent Treatment with Prolonged Exposure (COPE)
- Treatment as usual (Active Comparator): CBT for substance use disorder.
  Interventions: Behavioral: Concurrent Treatment with Prolonged Exposure (COPE)

INTERVENTIONS:
Behavioral: Concurrent Treatment with Prolonged Exposure (COPE) — 12 weeks of concurrent prolonged exposure treatment for PTSD combined with cognitive behavioral therapy for substance use disorders (alcohol or drugs).
  Other Names: Prolonged Exposure

SUMMARY:
In comparison to the general population, U.S. military and Veterans are at an increased risk for developing both substance use disorders (SUD) and Post Traumatic Stress Disorder (PTSD). Current research has shown that there is a high comorbidity of SUD and PTSD, and although there are a number of treatments for SUD and PTSD independently, there are very few effective methods to simultaneously treat both disorders. Because of this substantial gap in the treatment of both SUDs and PTSD, it has become essential to develop a combined treatment that would address and treat both disorders. Individuals, specifically U.S. military and Veterans, with SUD/PTSD have unique needs that require a specialized treatment approach. This designed approach would employ cognitive-behavioral therapy (CBT) to treat the SUD, in conjunction with Prolonged Exposure therapy to treat the PTSD. Prolonged Exposure (PE) is an empirically supported and evidence-based treatment that is currently regarded as the "gold standard" psychosocial treatment for PTSD. In combination with CBT, this treatment would address both disorders in hopes of reducing substance use and PTSD symptomatology.

DETAILED DESCRIPTION:
As a result of sustained operations in Afghanistan and Iraq, there are an increasing number of U.S. military personnel and Veterans at risk of developing both substance use disorders (SUDs) and Post Traumatic Stress Disorder (PTSD). If left untreated, individuals with SUDs and/or PTSD are at risk for other mental health problems (e.g., depression), suicidal ideation and attempts, physical health problems, reduced resiliency, lost productivity, and family/relationship impairment. While mental health services are in place for U.S. military personnel, substantial gaps in the treatment of co-occurring SUDs and PTSD exist and there is little scientific evidence available to guide the provision of care. The proposed study directly addresses this knowledge gap by testing the feasibility and preliminary efficacy of an integrative behavioral intervention for the treatment of co-occurring SUDs and PTSD modified for use among U.S. military personnel (including National Guard and Reservists) who have served in Operation Enduring Freedom and/or Operation Iraqi Freedom (OEF/OIF). The intervention, called "Concurrent Treatment with Prolonged exposure" or "COPE," represents a novel treatment that integrates cognitive-behavioral therapy for SUDs with prolonged exposure therapy for PTSD. In earlier studies with civilians, COPE has demonstrated efficacy in reducing alcohol and drug use severity, PTSD symptoms, and associated mental health problems (e.g., depression, anxiety). In this hybrid Stage Ib/Stage II study, we will (1) use a manualized, well-tolerated behavioral treatment for SUDs and PTSD (COPE); (2) employ a two-arm randomized between-groups experimental design (COPE versus a modified treatment-as usual (TAU); and (3) examine standardized, repeated dependent measures of clinical outcomes and process variables at 5 time points (pre-, mid-, and post-treatment; 3 and 6 month follow-up). The proposed project is directly responsive to the mission of the National Institute on Drug Abuse (NIDA) and the National Institute on Alcohol Abuse and Alcoholism (NIAAA) in that it seeks to enhance and accelerate research on the prevention and treatment of alcohol and drug use disorders (including illicit and prescription drugs) and comorbid conditions (e.g., PTSD, depression, sleep disturbances, HIV risk behaviors). The findings of this study will provide empirical evidence to inform policies and programs to better serve the needs of U.S. military personnel, Veterans, and their families.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active-duty OIF/OEF military personnel and separated OIF/OEF veterans ages 18-65.
* Diagnosis of PTSD determined by a clinician-administered study interview.

Exclusion Criteria:

* Current bipolar disorder or other psychotic disorder (as determined by the evaluator conducting the patient interview and medical record review)
* subjects with a current eating disorder or with dissociative identity disorder
* currently in ongoing therapy for SUDs or PTSD, who are not willing to discontinue these therapies for the duration of the trial
* recently prescribed maintenance anxiolytic, antidepressant, or mood stabilizing medications (must be stabilized for four weeks on meds before entry into study)
* Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudie E Back, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szafranski DD, Snead A, Allan NP, Gros DF, Killeen T, Flanagan J, Pericot-Valverde I, Back SE. Integrated, exposure-based treatment for PTSD and comorbid substance use disorders: Predictors of treatment dropout. Addict Behav. 2017 Oct;73:30-35. doi: 10.1016/j.addbeh.2017.04.005. Epub 2017 Apr 4. PMID 28460246
- [Background] Mills AC, Badour CL, Korte KJ, Killeen TK, Henschel AV, Back SE. Integrated Treatment of PTSD and Substance Use Disorders: Examination of Imaginal Exposure Length. J Trauma Stress. 2017 Apr;30(2):166-172. doi: 10.1002/jts.22175. Epub 2017 Mar 22. PMID 28329434
- [Background] Korte KJ, Bountress KE, Tomko RL, Killeen T, Moran-Santa Maria M, Back SE. Integrated Treatment of PTSD and Substance Use Disorders: The Mediating Role of PTSD Improvement in the Reduction of Depression. J Clin Med. 2017 Jan 13;6(1):9. doi: 10.3390/jcm6010009. PMID 28098747
- [Background] Lancaster CL, Gros DF, Mullarkey MC, Badour CL, Killeen TK, Brady KT, Back SE. Does trauma-focused exposure therapy exacerbate symptoms among patients with comorbid PTSD and substance use disorders? Behav Cogn Psychother. 2020 Jan;48(1):38-53. doi: 10.1017/S1352465819000304. Epub 2019 Apr 23. PMID 31010449
- [Result] Back SE, Killeen T, Badour CL, Flanagan JC, Allan NP, Ana ES, Lozano B, Korte KJ, Foa EB, Brady KT. Concurrent treatment of substance use disorders and PTSD using prolonged exposure: A randomized clinical trial in military veterans. Addict Behav. 2019 Mar;90:369-377. doi: 10.1016/j.addbeh.2018.11.032. Epub 2018 Nov 27. PMID 30529244
- [Result] Badour CL, Flanagan JC, Gros DF, Killeen T, Pericot-Valverde I, Korte KJ, Allan NP, Back SE. Habituation of distress and craving during treatment as predictors of change in PTSD symptoms and substance use severity. J Consult Clin Psychol. 2017 Mar;85(3):274-281. doi: 10.1037/ccp0000180. PMID 28221062

RESULTS

PARTICIPANT FLOW:
Groups:
- COPE Therapy: Combined prolonged exposure therapy for PTSD with cognitive behavioral therapy for substance use.
  Concurrent Treatment with Prolonged Exposure (COPE): 12 weeks of concurrent prolonged exposure treatment for PTSD combined with cognitive behavioral therapy for substance use disorders (alcohol or drugs).
- Treatment as Usual: Current standard treatment available through the Department of Veteran's Affairs.
  Concurrent Treatment with Prolonged Exposure (COPE): 12 weeks of concurrent prolonged exposure treatment for PTSD combined with cognitive behavioral therapy for substance use disorders (alcohol or drugs).
Period: Overall Study
Arm/Group | COPE Therapy | Treatment as Usual
Started | 54 | 27
Completed | 29 | 13
Not Completed | 25 | 14

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual: Relapse Prevention (RP) for substance use disorders.
  Included 12 sessions of RP matched for time.
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | COPE Therapy | Total
Number analyzed (Participants) | 27 | 54 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants were asked their age at baseline visit using a demographic form.
  years | 41.9 (10.3) | 39.7 (11.0) | 40.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 23 | 50 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 26 | 52 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 16 | 30
  White | 12 | 37 | 49
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 54 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-traumatic Stress Disorder Symptomatology
Description: The hypothesis is that COPE will significantly exceed the treatment as usual control group in reducing Change in Post-traumatic Stress Disorder symptoms as measured by a reduction of 25 points or more in scores for the Clinician Administered Post-traumatic Stress Disorder Scale (CAPS).
  A lower Clinician Administered Post-traumatic Stress Disorder Scale and Post-traumatic Stress Disorder Checklist score would indicate less severe Post-traumatic Stress Disorder/better outcomes.
  A negative sign in front of a number represents a decrease in score and better/positive outcomes. A greater decrease in a score represents greater improvement in symptoms (more positive outcomes).
  Clinician Administered Post-traumatic Stress Disorder Scale (CAPS): scores range 0-136 0-19: asymptomatic/few symptoms 20-39: mild PTSD/subthreshold 40-59: moderate PTSD/threshold 60-79: severe PTSD symptoms
  ≥80: extreme PTSD symptoms
  Post-traumatic Stress Disorder Checklist: score range 17-85.
Time Frame: Following 12 weeks of therapy.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | COPE Therapy | Treatment as Usual
Number analyzed (Participants) | 54 | 27
score on a scale
  Clinician Administered PTSD Sore | -51.2 [-59.7 to -42.8] | -35.9 [-48.8 to -23]
  The PTSD Checklist for DSM-5 PTSD Diagnosis | -22.3 [-29.3 to -15.3] | -10.9 [-18 to -3.9]

2. Primary Outcome: Drinks Per Drinking Day
Description: Number of standard drinks reported during drinking day
Time Frame: Following 12 weeks of therapy.
Measure: Mean (Standard Deviation); unit: Number of drinks per drinking day
Arm/Group | COPE Therapy | Treatment as Usual
Number analyzed (Participants) | 54 | 27
Number of drinks per drinking day | 4.6 (3.6) | 5.0 (4.1)

3. Primary Outcome: Post-traumatic Stress Disorder Symptomatology
Description: Score of PTSD from Clinician Administered PTSD Scale (CAPS) and self-administered PTSD Checklist for DSM-5 PTSD Diagnosis (PCL-5).
  Lower scores on CAPS and PCL would indicate less severe PTSD. A lower Clinician Administered Post-traumatic Stress Disorder Scale and Post-traumatic Stress Disorder Checklist score would indicate less severe Post-traumatic Stress Disorder/better outcomes.
  A negative sign in front of a number represents a decrease in score and better/positive outcomes. A greater decrease in a score represents greater improvement in symptoms (more positive outcomes).
  Clinician Administered Post-traumatic Stress Disorder Scale (CAPS): scores range 0-136 0-19: asymptomatic/few symptoms 20-39: mild PTSD/subthreshold 40-59: moderate PTSD/threshold 60-79: severe PTSD symptoms
  ≥80: extreme PTSD symptoms
  Post-traumatic Stress Disorder Checklist: score range 17-85.
Time Frame: Following 12 weeks of therapy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COPE Therapy | Treatment as Usual
Number analyzed (Participants) | 54 | 27
score on a scale
  Clinician Administered PTSD Scale (CAPS) | 27.2 (19.4) | 49.7 (25.3)
  PTSD Checklist for DSM-4 PTSD Diagnosis (PCL-5) | 37.6 (17.2) | 53.1 (14.5)

4. Primary Outcome: Clinician Administered PTSD Scale Itemized Scores
Description: Clinician Administered PTSD Scale Itemized Scores Within the assessment there are 20 symptoms of PTSD, each with an individual score.
  A lower score would represent a better outcome (ie less severe symptom). The three itemized symptoms listed below represent hallmark traits/symptoms of PTSD.
  Overall score range 0-136 Reexperiencing Symptoms range 0-40 Avoidance/Numbing range 0-56 Hyperarousal range 0-40
Time Frame: After 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COPE Therapy | Treatment as Usual
Number analyzed (Participants) | 54 | 27
score on a scale
  Clinician Administered PTSD Scale- Re-experiencing | 5.6 (7.1) | 14.6 (10.7)
  Clinician Admin PTSD Scale - Avoidance/Numbing | 10.8 (9.7) | 24 (13.4)
  Clinician Administered PTSD Scale - Hyperarousal | 11.7 (8.2) | 19.1 (6.0)

5. Secondary Outcome: Number of Participants Who Report Abstinence
Description: The hypothesis is that COPE will significantly exceed the treatment as usual control group in reducing substance use as measured by decreases in percent days using and increased abstinence rates.
Time Frame: Following 12 weeks of therapy.
Population: Reported rate of abstinence
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | COPE Therapy
Number analyzed (Participants) | 27 | 54
Participants | 7 | 22

6. Secondary Outcome: Beck Depression Index
Description: Measure of depression. A lower score would indicate less severe depression. Scores range 0-30
Time Frame: Following 12 weeks of therapy.
Measure: Mean (Standard Deviation); unit: units on a scale (BDI)
Arm/Group | COPE Therapy | Treatment as Usual
Number analyzed (Participants) | 54 | 27
units on a scale (BDI) | 13 (11) | 19.4 (12.3)

ADVERSE EVENTS:
Arm/Group | COPE Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/54 | 1/27
Other Adverse Events (participants affected / at risk) | 0/54 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COPE Therapy (N=54) | Treatment as Usual (N=27)
Attempted suicide (Psychiatric disorders) | 0 (0) | 1 (1)
hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalized for suicidal ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No